CLINICAL TRIAL: NCT05210283
Title: CORRECT-MRD II: Second Colorectal Cancer Clinical Validation Study to Predict Recurrence Using a Circulating Tumor DNA Assay to Detect Minimal Residual Disease
Brief Title: CORRECT Study of Minimal Residual Disease Detection in Colorectal Cancer
Acronym: MRD
Status: Active, not recruiting | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Collaborators: NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Other Study IDs: 16-002
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
Keywords: Colorectal; ctDNA
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Stage ll or lll: Patients with stage ll or lll colorectal cancer
  Interventions: Device: MRD

INTERVENTIONS:
Device: MRD — ctDNA MRD test

SUMMARY:
The CORRECT - MRD II study will prospectively enroll patients who have undergone complete surgical resection for stage II or III colorectal cancer. Maximum duration of participant participation is up to seven years from enrollment to study completion with up to five years of active follow up and up to two years of clinical (passive) follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of carcinoma of the colon or rectum (patients with lymphomatous, sarcomatous, or neuroendocrine features are not eligible).
2. Post complete surgical resection of CRC, with last surgery occurring within 180 days prior to enrollment are eligible if all of the following conditions are met:

   1. in the opinion of the surgeon, all grossly visible tumor was completely resected ("curative resection") and
   2. histologic evaluation by the pathologist confirms the margins of the resected specimens are not involved by malignant cells.

   i. Patients with T4 tumors that have involved an adjacent structure (e.g., bladder, small intestine, ovary, etc.) by direct extension from the primary tumor must have had all or a portion of the adjacent structure removed en bloc with the primary tumor and local radiation therapy will not be utilized.
3. Pathologic stage II or III
4. ECOG performance status ≤ 2 (0, 1 or 2).
5. Able to understand and provide informed consent.
6. Willing and able to comply with the study requirements, which includes the collection of approximately 43mL of blood for each research blood draw.

Exclusion Criteria:

1. Initiated adjuvant therapy for current CRC diagnosis (note: prior neoadjuvant therapy acceptable).
2. Pregnant or breastfeeding at time of enrollment.
3. Prior history of any invasive cancer (including CRC) within the past 3 years prior to informed consent, with the exception of non-melanoma skin cancer. Patients with a prior history of noninvasive (in situ) carcinomas may participate after definitive treatment.
4. Prior transplant history:

   1. Prior allogeneic hematopoietic stem cell transplant at any time.
   2. Prior solid organ transplant within the last 2 years prior to enrollment.
5. Multiple cancer diagnoses: Synchronous or asynchronous diagnoses (or suspicion) of multiple primary cancers at the time of eligibility screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who have undergone surgery for stage II or III colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 1017 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
To validate the association of circulating tumor DNA (ctDNA) with recurrence-free interval (RFI). | 7 years

SECONDARY OUTCOMES:
To assess the sensitivity and specificity of ctDNA positivity for subsequent clinical recurrence. | 7 years
To assess the contribution of ctDNA on RFI, independent of clinicopathological risk features and other biomarkers | 7 years
To assess time from positive ctDNA to clinical recurrence | 7 years

CONTACTS AND LOCATIONS:
Locations (32):
- United States (28):
  - Facey Medical Group - Mission Hills - Endoscopy Center & Gastroenterology, Mission Hills, California
  - Torrance Memorial Hunt Cancer Institute, Torrance, California
  - University of Florida Division of Hematology & Oncology, Gainesville, Florida
  - Mount Sinai Medical - Comprehensive Cancer Center, Miami Beach, Florida
  - Mid Florida Cancer Centers, Orange City, Florida
  - Edward Cancer Center, Elmhurst, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Mercy Medical Center, Cedar Rapids, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - MedStar Georgetown Cancer Institute at MedStar Georgetown University Hospital, Baltimore, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - University of Maryland St. Joseph Medical Center, Towson, Maryland
  - Metro Minnesota Community Oncology Consortium (MMCORC), Saint Louis Park, Minnesota
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Columbus NCORP, Columbus, Ohio
  - Interstate Medical Office Central, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Reading Hospital Hematology Oncology, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan York Cancer Center, York, Pennsylvania
  - Primsa Health Cancer Institute, Greenville, South Carolina
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - Ballad Health Cancer Center, Kingsport, Tennessee
  - Marshfield Medical Center Weston, Weston, Wisconsin
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health - Glen Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after deidentification. This may include test, tables, figured, and appendices. The study protocol, statistical analysis plan (when applicable), informed consent form (when applicable). May not be reproduced nor disseminated outside of Exact Sciences without permission and the clinical study report (when applicable) will also be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available from 2 years and ending 4 years after publication
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary Institutional Review Board (IRB)/Institutional Ethics Committee (IEC) approvals or waivers as applicable to conduct research.